CLINICAL TRIAL: NCT01484431
Title: A Multiple Ascending Dose Study of Tadalafil to Assess the Pharmacokinetics and Safety in a Pediatric Population With Pulmonary Arterial Hypertension
Brief Title: A Pharmacokinetics Study for Pediatric Participants With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12917; H6D-MC-LVIG (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Tadalafil; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tadalafil (Experimental): Light Weight <25 kg Period 1: 2 milligram (mg) or 4 mg tadalafil administered once daily (QD) in oral suspension formulation for 5 weeks then 8 mg,10 mg,15 mg or 20 mg tadalafil was administered QD in oral suspension formulation for 5 weeks.
  Middle Weight: 25 kg to <40 kg Period 1: 5 mg tadalafil tablet administered QD for 5 weeks then 10 mg, 15 mg or 20 mg tablet tadalafil administered QD for 5 weeks.
  Heavy: ≥40 kg Period 1: 10 mg tadalafil tablet administered QD for 5 weeks then 20 mg or 40 mg tablet tadalafil administered QD for 5 weeks.
  Interventions: Drug: Tadalafil- Tablet or Oral suspension

INTERVENTIONS:
Drug: Tadalafil- Tablet or Oral suspension — Tadalafil Tablets administered orally. Tadalafil Oral suspension: An aqueous, ready-to-use suspension for oral administration.
  Other Names: LY450190

SUMMARY:
The purpose of this study is to see how much study drug is in the blood of children with pulmonary arterial hypertension (PAH) after dosing to establish the correct dose for further clinical research.

DETAILED DESCRIPTION:
During Period I, tadalafil will be administered orally, once daily, at a low dose for approximately 5 weeks followed by a high dose for approximately 5 weeks. Dose levels are calculated based on body weight cohorts. Heavy weight cohort >=40 kg, middle weight cohort >=25 kg to <40 kg. Light weight cohort<25 kg. Participants who complete Period 1 may continue taking tadalafil in Period 2 for at least 2 years. Starting dose will not exceed the maximum weight range dose established in Period 1 and after the first 3 months of Period 2, the dose may be adjusted based on available safety and efficacy information.

ELIGIBILITY:
Inclusion Criteria:

* Currently have a diagnosis of PAH that is either:

  * idiopathic (including hereditary), related to collagen vascular disease, related to anorexigen use, associated with surgical repair, of at least 6 month duration, of a congenital systemic to pulmonary shunt (for example, atrial septal defect, ventricular septal defect, patent ductus arteriosus).
* Have a history of the diagnosis of PAH established by a resting mean pulmonary artery pressure ≥25 mm Hg, pulmonary artery wedge pressure ≤15 mm Hg, and a pulmonary vascular resistance (PVR) ≥3 Wood units via right heart catheterization. In the event that a pulmonary artery wedge pressure is unable to be obtained during right heart catheterization, participants with a left ventricular end diastolic pressure <15 mm Hg, with normal left heart function, and absence of mitral stenosis on echocardiography can be eligible for enrollment
* Have a World Health Organization (WHO) functional class value of I, II or III at the time of enrollment

Exclusion Criteria:

* Have pulmonary hypertension related to conditions other than specified above, including but not limited to chronic thromboembolic disease, portal pulmonary hypertension, left-sided heart disease or lung disease and hypoxia
* History of left-sided heart disease, including any of the following:

  * clinically significant (pulmonary artery occlusion pressure [PAOP] 15 to 18 mm Hg) aortic or mitral valve disease (that is, aortic stenosis, aortic insufficiency, mitral stenosis, moderate or greater mitral regurgitation)
  * pericardial constriction
  * restrictive or congestive cardiomyopathy
  * left ventricular ejection fraction <40% by multigated radionucleotide angiogram (MUGA), angiography, or echocardiography
  * left ventricular shortening fraction <22% by echocardiography
  * life-threatening cardiac arrhythmias
  * symptomatic coronary artery disease within 5 years of study entry as determined by the physician
* History of atrial septostomy or Potts Shunt within 3 months before administration of study drug
* Unrepaired congenital heart disease

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (5):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's Heathcare of Atlanta, Inc. at Egleston, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomsbury, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: • Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Ferguson-Sells L, Velez de Mendizabal N, Li B, Small D. Population Pharmacokinetics of Tadalafil in Pediatric Patients with Pulmonary Arterial Hypertension: A Combined Adult/Pediatric Model. Clin Pharmacokinet. 2022 Feb;61(2):249-262. doi: 10.1007/s40262-021-01052-8. Epub 2021 Aug 11. PMID 34379314
- See also: Click here for more information about this study: A Pharmacokinetics Study for Pediatric Participants With Pulmonary Arterial Hypertension (PAH) — https://www.lillytrialguide.com/en-US/studies/pediatric-pulmonary-arterial-hypertension/LVIG#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol, the summary was based on weight cohorts.
Pre-assignment Details: This study contains 2 periods: Pharmacokinetics(PK)/safety Period 1 and an open-label safety extension Period 2. Period 1 is approximately 10 weeks (that is, approximately 5 consecutive weeks for each dose [low and high]). Period 2 is at least 2 years after participating in Period 1.
Groups:
- Light Weight <25 kg: Period 1: 2 milligram (mg) or 4 mg tadalafil administered once daily (QD) in oral suspension formulation for 5 weeks then 8 mg,10 mg,15 mg or 20 mg tadalafil was administered QD in oral suspension formulation for 5 weeks.
  Period 2: Open Label Extension for 2 years.
  7 mg, 8 mg, 15 mg or 20 mg tadalafil administered once daily (QD) in oral suspension formulation.
- Middle Weight: 25 kg to <40 kg: Period 1: 5 mg tadalafil tablet administered QD for 5 weeks then 10 mg, 15 mg or 20 mg tablet tadalafil administered QD for 5 weeks.
  Period 2: Open Label Extension for 2 years.
  7.5 mg, 10 mg, 15 mg or 20 mg tadalafil administered once daily (QD) in oral tablet.
- Heavy Weight: ≥40 kg: Period 1: 10 mg tadalafil tablet administered QD for 5 weeks then 20 mg or 40 mg tablet tadalafil administered QD for 5 weeks.
  Period 2: Open Label Extension for 2 years.
  15 mg, 20 mg or 40 mg tadalafil administered once daily (QD) in oral tablet.
Period: Period 1: Low Dose
Arm/Group | Light Weight <25 kg | Middle Weight: 25 kg to <40 kg | Heavy Weight: ≥40 kg
Started | 6 | 7 | 6
Received 2 mg | 1 | 0 | 0
Received 4 mg | 5 | 0 | 0
Received 5 mg | 0 | 7 | 0
Received 10 mg | 0 | 0 | 6
Completed | 6 | 7 | 6
Not Completed | 0 | 0 | 0
Period: Period 1: High Dose
Arm/Group | Light Weight <25 kg | Middle Weight: 25 kg to <40 kg | Heavy Weight: ≥40 kg
Started | 6 | 7 | 6
Received 8 mg | 1 | 0 | 0
Received 10 mg | 1 | 1 | 0
Received 15 mg | 1 | 1 | 0
Received 20 mg | 3 | 5 | 1
Received 40 mg | 0 | 0 | 5
Completed | 6 | 6 | 6
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: Period 2
Arm/Group | Light Weight <25 kg | Middle Weight: 25 kg to <40 kg | Heavy Weight: ≥40 kg
Started | 6 | 6 | 6
Received 7 mg | 1 | 0 | 0
Received 7.5 mg | 0 | 2 | 0
Received 8 mg | 1 | 0 | 0
Received 10 mg | 0 | 1 | 0
Received 15 mg | 1 | 2 | 1
Received 20 mg | 3 | 1 | 4
Received 40 mg | 0 | 0 | 1
Completed | 5 | 5 | 4
Not Completed | 1 | 1 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Non-Compliance with Study Drug | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug. Participants were first administered a low dose to explore PK of tadalafil and determine a high dose within the weight cohort. Per protocol, the summary was based on weight cohorts.
Groups:
- Light Weight: <25 kg: Period 1: 2 milligram (mg) or 4 mg tadalafil administered once daily (QD) in oral suspension formulation for 5 weeks then 8 mg,10 mg,15 mg or 20 mg tadalafil was administered QD in oral suspension formulation for 5 weeks.
- Middle Weight: 25 kg to <40 kg: Period 1: 5 mg tadalafil tablet administered QD for 5 weeks then 10 mg, 15 mg or 20 mg tablet tadalafil administered QD for 5 weeks.
- Heavy Weight: ≥40 kg: Period 1: 10 mg tadalafil tablet administered QD for 5 weeks then 20 mg or 40 mg tablet tadalafil administered QD for 5 weeks.
- Total: Total of all reporting groups
Arm/Group | Light Weight: <25 kg | Middle Weight: 25 kg to <40 kg | Heavy Weight: ≥40 kg | Total
Number analyzed (Participants) | 6 | 7 | 6 | 19
Age, Continuous [Mean (Full Range); unit: years] | 5.00 [2.5 to 8.0] | 10.91 [7.3 to 17.9] | 14.45 [11.3 to 17.6] | 10.16 [2.5 to 17.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 13
  Male | 2 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 4 | 5 | 5 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 1 | 1 | 5
  United States | 1 | 0 | 1 | 2
  Poland | 1 | 2 | 2 | 5
  United Kingdom | 0 | 3 | 0 | 3
  France | 0 | 1 | 1 | 2
  Spain | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Population Pharmacokinetics: Area Under the Concentration Curve Versus Time at a Dosing Interval at Steady State (AUCtau) for Tadalafil
Description: Population Pharmacokinetics: Area Under the Concentration Curve Versus Time at a Dosing Interval at Steady State (AUCtau) for Tadalafil.
  The measure of dispersion reported is 90% Prediction Intervals and not Confidence Intervals.
Time Frame: Period 1: Pre Dose and 2, 4, 8, 12, and 24 Hours Post Dose on Days 1, 14 and 49; with single dose measures on Day 1 and steady-state measurements on Days 14 and 49
Population: All participants who received at least one dose of study drug and had evaluable PK data including all dose levels on Day 1, 14 and 49. Per protocol, the summary reflects potential exposure of the high dose within each weight cohort
Measure: Median (90% Confidence Interval); unit: nanograms* hour per milliliter(ng*hr/mL)
Groups:
- 20 mg Light Weight: <25 kg: 20 mg tadalafil administered QD in oral suspension formulation.
- 20 mg Middle Weight: 25 kg to <40 kg: 20 mg tablet tadalafil administered QD.
- 40 mg Heavy Weight: ≥40 kg: 40 mg tablet tadalafil administered QD.
Arm/Group | 20 mg Light Weight: <25 kg | 20 mg Middle Weight: 25 kg to <40 kg | 40 mg Heavy Weight: ≥40 kg
Number analyzed (Participants) | 6 | 7 | 6
nanograms* hour per milliliter(ng*hr/mL)
  Not Taking Bosentan | 8170 [3850 to 16700] | 8390 [4130 to 18400] | 15200 [6980 to 31100]
  Taking Concomitant Bosentan | 4550 [2170 to 9450] | 5000 [2440 to 10600] | 8990 [4270 to 19500]

2. Primary Outcome: Population Pharmacokinetics: Average Concentration (Cmean,ss) of for Tadalafil at Steady-State.
Description: Population Pharmacokinetics: Average Concentration (Cmean,ss) of for tadalafil at steady-state.
  The measure of dispersion reported is 90% Prediction Intervals and not Confidence Intervals.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Groups:
- 20 mg Light Weight <25 kg: 20 mg tadalafil administered QD in oral suspension formulation.
Arm/Group | 20 mg Light Weight <25 kg | 20 mg Middle Weight: 25 kg to <40 kg | 40 mg Heavy Weight: ≥40 kg
Number analyzed (Participants) | 6 | 7 | 6
nanograms per milliliter (ng/mL)
  Not Taking Bosentan | 340 [161 to 694] | 350 [172 to 767] | 633 [291 to 1300]
  Taking Concomitant Bosentan | 190 [90.4 to 394] | 209 [102 to 440] | 375 [178 to 815]

3. Secondary Outcome: Percentage of Participants With Clinical Worsening
Description: Clinical worsening was defined as any of the following: death, lung or heart transplantation, atrial septostomy or Potts' shunt, hospitalization for Pulmonary Arterial Hypertension (PAH) progression, new onset syncope, initiation of new PAH therapy (including increase in the dose of existing PAH specific concomitant therapy, such as endothelin receptor agonist or beraprost medication), or increase of 1 or more in World Health Organization(WHO) Functional Class (except for participants already in Class IV; only for participants unable to perform the 6 minute walk (6MW) test; worsening of WHO functional class by 1 or more for participants who can perform a 6 minute walk (6MW) test and who have a decrease of ≥ 20% in the 6 minute walk distance (for those participants who are ≥6 years of age).
Time Frame: Baseline Up to 27 Months
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Light Weight <25 kg | Middle Weight: 25 kg to <40 kg | Heavy Weight: ≥40 kg
Number analyzed (Participants) | 6 | 7 | 6
percentage of participants | 50.00 | 28.57 | 33.33

4. Secondary Outcome: Number of Participants With Palatability of the Tadalafil Suspension
Description: The Taste Assessment Questionnaire (TAQ) questions were:
  TAQRES1: Please rate the bitterness level. TAQRES2: Please rate the sweetness level. TAQRES3: Please rate the aftertaste. TAQRES4: Please rate the overall acceptability of the taste for daily use.
Time Frame: Day 35 (high dose)
Population: Participants who received at least one oral suspension dose of study drug in the Light-weight cohort (≥2 years of age). Per protocol, palatability of the tadalafil suspension was evaluated in the Light-weight cohort only.
Measure: Count of Participants; unit: Participants
Arm/Group | Light Weight: <25 kg
Number analyzed (Participants) | 3
Participants
  TAQRES1: Extremely bitter | 0
  TAQRES1: Very bitter | 0
  TAQRES1: Moderately bitter | 0
  TAQRES1: Slightly bitter | 0
  TAQRES1: Not bitter | 3
  TAQRES2: Extremely sweet | 1
  TAQRES2: Very sweet | 0
  TAQRES2: Moderately sweet | 1
  TAQRES2: Slightly sweet | 1
  TAQRES2: Not sweet | 0
  TAQRES3: Extreme aftertaste | 0
  TAQRES3: Strong aftertaste | 1
  TAQRES3: Moderate aftertaste | 0
  TAQRES3:Slight aftertaste | 0
  TAQRES3:No aftertaste | 2
  TAQRES4: Not acceptable | 0
  TAQRES4: Slightly acceptable | 0
  TAQRES4: Acceptable | 2
  TAQRES4: Very acceptable | 1

ADVERSE EVENTS:
Time Frame: Up To 27 Months
Description: All participants who received at least one dose of study drug. Participants were first administered a low dose to explore PK of tadalafil and determine a high dose within the weight cohort. Per protocol, the summary was based on weight cohorts. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Light Weight: <25 kg: Period 1: 2 milligram (mg) or 4 mg tadalafil administered once daily (QD) in oral suspension formulation for 5 weeks then 8 mg,10 mg,15 mg or 20 mg tadalafil was administered QD in oral suspension formulation for 5 weeks.
  Period 2: Open Label Extension for 2 years.
  7 mg, 8 mg, 15 mg or 20 mg tadalafil administered once daily (QD) in oral suspension formulation.
- Middle Weight: 25 kg to <40 kg: Period 1: 5 mg tadalafil tablet administered QD for 5 weeks then 10 mg, 15 mg or 20 mg tablet tadalafil administered QD for 5 weeks.
  Period 2: Open Label Extension for 2 years.
  7.5 mg, 10 mg, 15 mg or 20 mg tadalafil administered once daily (QD) in oral tablet.
  .
Arm/Group | Light Weight: <25 kg | Middle Weight: 25 kg to <40 kg | Heavy Weight: ≥40 kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/7 | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/7 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Light Weight: <25 kg (N=6) | Middle Weight: 25 kg to <40 kg (N=7) | Heavy Weight: ≥40 kg (N=6)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/4 (0) | 0/5 (0) | 1/4 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Light Weight: <25 kg (N=6) | Middle Weight: 25 kg to <40 kg (N=7) | Heavy Weight: ≥40 kg (N=6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (4)
Pyrexia (General disorders) | 2 (7) | 1 (1) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 1 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (5) | 1 (1) | 2 (7)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (5)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cytogenetic analysis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Exercise test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/4 (0) | 0/5 (0) | 1/4 (1)
Menorrhagia (Reproductive system and breast disorders) | 0/4 (0) | 0/5 (0) | 1/4 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0/4 (0) | 0/5 (0) | 1/4 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (4) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasodilatation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-06-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT01484431/Prot_000.pdf
  • Statistical Analysis Plan (2012-08-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT01484431/SAP_001.pdf